CLINICAL TRIAL: NCT04314258
Title: Randomized Clinical Study Investigating the Effect of Moringa Oleifera Infusion on Bioclinical Parameters of Health
Brief Title: Effect of Moringa Oleifera Infusion on Health
Acronym: MOI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Mauritius (Other)
Responsible Party: Principal Investigator, MChanSun, Associate Professor, University of Mauritius
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UOM002
Record Dates: First submitted 2020-02-18; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: This randomized clinical study will consist of two parallel groups with a crossover design.
  There will be two arms as follows:
  1. Intervention group [Drinking Moringa tea]
  2. Control group [Drinking plain water].
  Computer-generated random numbers will be used for simple randomization of subjects to either the experimental or control group.
  With the cross over design, there will be two phases with an interchange of the groups during Phase 1 and 2 as follows:
  Four-week Phase 1 - Group A drinking Moringa tea v/s Group B drinking plain water One-week washout Four-week Phase 2 - Group A drinking plain water v/s Group B drinking Moringa tea
Who Masked: Outcomes Assessor
Masking Description: A coding system will be used whereby each subject will be attributed a code upon signing the consent form. Only the Principal Investigator assisted by a second investigator will have access to the name-code list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drinking Moringa oleifera tea (Experimental): The experimental group will drink twice daily 2 tea bags of Moringa oleifera tea (Kanhye brand) infused in 200 ml of hot water (during 5 minutes) for a period of 4 weeks. The locally available Moringa tea with the international certification by ECOCERT France will be used in this study.
  Interventions: Dietary Supplement: Moringa oleifera tea
- Drinking plain water (No Intervention): The control group will receive instructions to consume 200 ml of plain water twice daily for a period of 4 weeks.

INTERVENTIONS:
Dietary Supplement: Moringa oleifera tea — 4 grams of Moringa oleifera tea twice daily
  Arms: Drinking Moringa oleifera tea

SUMMARY:
The study aims at investigating the effects of the consumption of Moringa oleifera Lam leaves on biomedical markers of health among healthy individuals who are hyperglycaemic with a fasting blood glucose equal or greater than 5.5mmol/L.

The main objectives are as follows:

1. To determine the effect of consuming 4 grams of Moringa oleifera Lam leaves infused in 200 ml of hot water twice daily on blood glucose level [BSc (Hons) Medical Science Student].
2. To assess the effect of consuming 4 grams of Moringa oleifera Lam leaves infused in 200 ml of hot water twice daily on plasma lipids level [Master of Public Health Students].
3. To compare the effect of the Moringa tea consumption on lipid profiles of both healthy and hyperglycemic participants [Master of Public Health Students].
4. To evaluate the effects of Moringa oleifera Lam leaves on blood anti-oxidant status [BSc (Hons) Nutritional Sciences Student].

The research work will consist of (1) Experimental intervention: The experimental group will drink Moringa tea; (2) Survey questionnaire, (3) Anthropometric measurements, (4) Blood pressure determination and (5) Blood collections at 15-day intervals during 9 weeks. The blood tests to be performed are as follows: Glucose, HbA1C, Uric acid, C-Protein reactive, Lipid Profile (Total Cholesterol, HDL Cholesterol, Triglycerides), and blood antioxidants (superoxide dismutase, glutathione peroxidase, total blood anti-oxidant capacity).

DETAILED DESCRIPTION:
Study population

120 participants to include 60 healthy individuals and 60 individuals who are hyperglycaemic with a fasting blood glucose equal or greater than 5.5mmol/L will be recruited by means of flyers, posters and mass email by the help of Staff Club of the UoM.

Experimental design

This research work will to be undertaken under the responsibility and coordination of the Applicant who is the Principal Investigator working with two Academic Supervisors for the supervision of the four student projects.

This randomized clinical study will consist of two parallel groups with a crossover design.

There will be two arms as follows for each group:

1. Intervention group [drinking Moringa tea] and
2. Control group [drinking plain water].

Computer-generated random numbers will be used for simple randomization of subjects to either the experimental or control (equal amount of water) groups. Half of the participants will be assigned to the experimental group and the other control (water) for the first 4 weeks during Phase 1.

The experimental group will be provided with Moringa tea bags and instructed to consume twice daily 2 tea bags (4 tea bags equivalent to 8 grams) of Moringa tea (Kanhye brand) infused in 200 ml of hot water (during 5 minutes) for a period of 4 weeks. The locally available Moringa tea with the international certification by ECOCERT France will be used in this study.

With the cross over design, there will be two phases for both healthy and hyperglycaemic groups with an interchange of the groups during Phase 1 and 2 as follows:

Four-week Phase 1 - Group A drinking Moringa tea v/s Group B drinking plain water One-week washout Four-week Phase 2 - Group A drinking plain water v/s Group B drinking Moringa tea

The duration of the clinical study will normally be nine weeks with possible extension of four weeks.

Outcome Measurements Baseline data collection Measurements of body weight and blood pressure will be performed. Anthropometric measurements will be taken for each subject: Weight will be measured using an electronic weighing machine, height will be measured using a stadiometer, waist circumference will be measured using a non-stretchable measuring tape. Blood pressure will be measured using a sphygmomanometer.

Blood samples will be drawn by Specialized Nursing Officers from right or left ante-cubital vein of participant after a 12-h overnight fast. Blood tests which will be performed are as follows: Glucose, Lipid profile [Triglycerides, Total Cholesterol and HDL Cholesterol levels (LDL Cholesterol being calculated)], Uric Acid, HbA1C, C-Reactive Protein (hs-CRP) and Blood anti-oxidants (superoxide dismutase, glutathione peroxidase, total blood anti-oxidant capacity).

Fortnight monitoring sessions All participants of the two groups will be monitored on a fortnight basis for body weight, height, waist circumference, blood pressure and specified blood tests. Food intake and physical exercise questionnaires will be collected from participants to determine confounding factors.

[The individual quantity of physical activity, in metabolic equivalent-minutes per week (MET-min/week), will be determined by using validated physical activity questionnaire].

Outcome Measurements Baseline data collection Measurements of body weight and blood pressure will be performed. Anthropometric measurements will be taken for each subject: Weight will be measured using an electronic weighing machine, height will be measured using a stadiometer, waist circumference will be measured using a non-stretchable measuring tape. Blood pressure will be measured using a sphygmomanometer.

Blood samples will be drawn by Specialized Nursing Officers from right or left ante-cubital vein of participant after a 12-h overnight fast. Blood tests which will be performed are as follows: Glucose, Lipid profile [Triglycerides, Total Cholesterol and HDL Cholesterol levels (LDL Cholesterol being calculated)], Uric Acid, HbA1C, C-Reactive Protein (hs-CRP) and Blood anti-oxidants (superoxide dismutase, glutathione peroxidase, total blood anti-oxidant capacity).

Fortnight monitoring sessions All participants of the two groups will be monitored on a fortnight basis for body weight, height, waist circumference, blood pressure and specified blood tests. Food intake and physical exercise questionnaires will be collected from participants to determine confounding factors.

[The individual quantity of physical activity, in metabolic equivalent-minutes per week (MET-min/week), will be determined by using validated physical activity questionnaire].

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal fasting plasma glucose levels
* Individuals with pre-diabetes condition newly diagnosed
* Individuals with dyslipidemia
* Type 2 Diabetes patients taking oral allopathic hypoglycemic agents

Exclusion Criteria:

* Pregnant women
* Smokers
* People with alcohol intake >2 standard drinks per day (in line with Bahorun et al. 2012)
* Patients with any complications of diabetes mellitus
* Patients on insulin therapy (in line with Leone et al. 2018)
* Patients with gastro-intestinal, hepatic, cardiovascular, renal or endocrine disorder (other than diabetes mellitus) which can interfere with the absorption, metabolism and excretion of Moringa leaves (in line with Bahorun et al. 2012)
* Patients on medication for diseases other than diabetes
* Persons taking botanical extracts
* People currently on a diet (in line with Ahmad et al. 2018)
* People having food allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose level | Eight weeks
  Change will be determined as the value at Day 29 with respect to Day 1 for Phase 1 (Four weeks) and for Phase 2 (four weeks)
Change in Low-density Lipoprotein (LDL) Cholesterol level | Eight weeks
  Change will be determined as the value at Day 29 with respect to Day 1 for Phase 1 (Four weeks) and for Phase 2 (four weeks)
Change in Triglyceride level | Eight weeks
  Change will be determined as the value at Day 29 with respect to Day 1 for Phase 1 (Four weeks) and for Phase 2 (four weeks)

SECONDARY OUTCOMES:
Change in levels of blood anti-oxidants | Eight weeks
  Levels of blood anti-oxidants (superoxide dismutase, glutathione peroxidase, total blood anti-oxidant capacity) will be monitored every fortnight during the 8-week clinical trial. C-Reactive Protein will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Marie CHAN SUN, PhD, Principal Investigator — University of Mauritius; Vidushi NEERGHEEN, PhD, Study Director — University of Mauritius; Abha JODHEEA-JUTTON, MD, Study Chair — University of Mauritius
Locations (1):
- University of Mauritius, Moka, Please Select, Mauritius

IPD SHARING:
Plan to Share IPD: Yes
CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2022-2025
Access Criteria: CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials.

REFERENCES:
- [Background] Bahorun T, Luximon-Ramma A, Neergheen-Bhujun VS, Gunness TK, Googoolye K, Auger C, Crozier A, Aruoma OI. The effect of black tea on risk factors of cardiovascular disease in a normal population. Prev Med. 2012 May;54 Suppl:S98-102. doi: 10.1016/j.ypmed.2011.12.009. Epub 2011 Dec 16. PMID 22198621
- [Background] Leone A, Bertoli S, Di Lello S, Bassoli A, Ravasenghi S, Borgonovo G, Forlani F, Battezzati A. Effect of Moringa oleifera Leaf Powder on Postprandial Blood Glucose Response: In Vivo Study on Saharawi People Living in Refugee Camps. Nutrients. 2018 Oct 12;10(10):1494. doi: 10.3390/nu10101494. PMID 30322091
- [Background] Ahmad J, Khan I, Johnson SK, Alam I, Din ZU. Effect of Incorporating Stevia and Moringa in Cookies on Postprandial Glycemia, Appetite, Palatability, and Gastrointestinal Well-Being. J Am Coll Nutr. 2018 Feb;37(2):133-139. doi: 10.1080/07315724.2017.1372821. Epub 2017 Dec 22. PMID 29272206
- [Background] Kumari, D. J. (2010) 'Hypoglycaemic Effect of Moringa Oleifera and Azadirachta Indica in Type 2 Diabetes Mellitus', The Bioscan, 5(2), p. 4.